CLINICAL TRIAL: NCT01861236
Title: Effectiveness and Safety of Firmagon® in Androgen Ablative Therapy of Advanced Hormone-dependent Prostate Carcinoma in Argentina
Acronym: FAST AR
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000036
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Advanced Hormone Dependent Prostate Cancer
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced Prostate Cancer: Advanced Prostate Cancer that receive Firmagon therapy in the context of usual clinical practice
  Interventions: Drug: Firmagon® (degarelix)

INTERVENTIONS:
Drug: Firmagon® (degarelix) — Monthly subcutaneous injections

SUMMARY:
Prospective, observational study to collect and analyze data on patients with advanced hormone dependent prostate cancer treated with Firmagon® according to routine medical practice in Argentina

ELIGIBILITY:
Inclusion Criteria:

* Advanced Prostate Cancer patients to be treated with Firmagon in the context of usual clinical practice
* Written informed consent

Exclusion Criteria:

* Contraindications to Firmagon
* Patients already on Firmagon therapy

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with Advanced Prostate Cancer that receive Firmagon therapy in the context of usual clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) failure rate (with failure defined as either prostate-specific antigen (PSA) failure, introduction of additional therapy related to prostate cancer, or death) | During 3 years treatment
  The PFS failure rate will be estimated with time to PFS failure as dependent and adjusting for disease stage at baseline, baseline PSA, baseline testosterone (if available) and baseline serum Alkaline Phosphatase (s-ALP, if available)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hospital de Trauma y Emergencia Dr Federico Abete, Ingeniero Pablo Nogués, Buenos Aires, Argentina